CLINICAL TRIAL: NCT07261787
Title: Duration of Surfactant Administration and Impact on Stabilisation of Vital Parameters in Very Preterm Neonates: 1 Minute Versus 5 Minutes - a Prospective Randomised-controlled Phase IV Trial - A Randomised Clinical Trial on Influence of Duration of Surfactant Administration on Stabilisation of Routine Monitoring Parameters and Cerebral Tissue Oxygen Saturation Monitoring in Preterm Neonates < 28 Weeks of Gestational Age
Brief Title: Duration of Surfactant Administration and Impact on Stabilisation of Vital Parameters in Very Preterm Neonates: 1 Minutes Versus 5 Minutes
Acronym: SurfStab I
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Christina Wolfsberger, MD, Priv.Doz. DDr., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SurfStab I Trial; 2025-522754-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Neonates and Preterm Infants; Infant Respiratory Distress Syndrome; Surfactant Deficiency Syndrome Neonatal; Surfactant; Cerebral Oxygenation; Cerebral Oxygen Saturation
Keywords: surfactant; surfactant administration; LISA; less-invasive surfactant administration; preterm neonates; cerebral oxygenation; near-infrared spectroscopy
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — poractant alfa; Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-Minute Administration ("1-min"-group) (Experimental): Infants receive poractant alfa (Curosurf®) administered via the LISA technique over 1 minute.
  Interventions: Drug: Poractant alfa (Curosurf®) - 1-minute administration
- 5-Minute Administration ("5-min"-group) (Experimental): Infants receive poractant alfa (Curosurf®) administered via the LISA technique over 5 minutes.
  Interventions: Drug: Poractant alfa (Curosurf®) - 5-minute administration

INTERVENTIONS:
Drug: Poractant alfa (Curosurf®) - 1-minute administration — Poractant alfa (Curosurf®, Chiesi Pharmaceuticals) administered intratracheally via the Less Invasive Surfactant Administration (LISA) technique over 1 minute.
  The surfactant is instilled manually through a thin catheter under direct laryngoscopy while the infant remains on continuous positive airway pressure (CPAP) and spontaneous breathing.
  Pre-specified criteria for aborting the LISA procedure are prolonged bradycardia (HR < 80 bpm) and/or arterial hypoxia (SpO2 < 80%) over 60 seconds during surfactant administration starting after the instillation of the LISA catheter. Data of included participants with discontinuation will be collected and analysed.
  Arms: 1-Minute Administration ("1-min"-group)
Drug: Poractant alfa (Curosurf®) - 5-minute administration — Poractant alfa (Curosurf®, Chiesi Pharmaceuticals) administered intratracheally via the Less Invasive Surfactant Administration (LISA) technique over 5 minute.
  The surfactant is instilled manually through a thin catheter under direct laryngoscopy while the infant remains on continuous positive airway pressure (CPAP) and spontaneous breathing.
  Pre-specified criteria for aborting the LISA procedure are prolonged bradycardia (HR < 80 bpm) and/or arterial hypoxia (SpO2 < 80%) over 60 seconds during surfactant administration starting after the instillation of the LISA catheter. Data of included participants with discontinuation will be collected and analysed.
  Arms: 5-Minute Administration ("5-min"-group)

SUMMARY:
Respiratory distress syndrome (RDS) is common in very preterm infants due to surfactant deficiency. Surfactant replacement therapy is lifesaving, and current guidelines recommend the less invasive surfactant administration (LISA) technique. However, the optimal duration of surfactant instillation during LISA has never been systematically evaluated. Rapid instillation may provoke transient hypoxia and bradycardia, while slower administration might improve physiological stability and cerebral oxygenation.

This randomised controlled trial investigates whether the duration of surfactant administration (1 minute versus 5 minutes) affects cerebral and systemic oxygen stability in extremely preterm neonates (< 28 weeks).

DETAILED DESCRIPTION:
The SurfStab I Trial is a single-centre, randomised, controlled, phase IV trial conducted at the Division of Neonatology, Department of Pediatrics and Adolescent Medicine, Medical University of Graz, Austria.

Infants born before 28 weeks of gestation and requiring surfactant therapy via the LISA technique will be randomised (1:1) to receive poractant alfa administered over either 1 minute or 5 minutes. The intervention duration represents two clinically accepted timeframes within current guideline recommendations.

Cerebral oxygenation will be monitored continuously using near-infrared spectroscopy (NIRS) from 5 minutes before to 3 hours after the procedure. The primary outcome is the maximal change in cerebral regional tissue oxygen saturation (crSO₂) from baseline (=5 minutes before starting the LISA procedure [insertion of the LISA catheter]) till 15 minutes after the LISA procedure (=removal of the LISA catheter). Secondary outcomes include changes in peripheral oxygen saturation (SpO₂), heart rate (HR), mean arterial blood pressure (MABP), frequency and duration of hypoxic or bradycardic episodes, and the need for repeated surfactant administration or invasive ventilation.

The total sample size is 76 infants (38 per arm). The study will provide evidence on whether slower surfactant administration improves physiological stability and cerebral oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonate <28+0 weeks (gestational age up to 27 weeks and 6 days)
* Indication of surfactant administration via the LISA method
* Postnatal age < 72 hours

Exclusion Criteria:

* Invasive ventilation, indication of INSURE procedure
* Severe pulmonary or cardiac malformation affecting oxygenation or congenital cerebral malformation
* Preexisiting diagnose of any IVH > grade 2 or PVH.

Ages: 0 Months to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral oxygenation (crSO₂) during and after LISA | From baseline (= 5min before insertion of the LISA catheter) till 15 minutes after removal of the thin catheter
  The primary outcome measure will be the maximum change of crSO2 from baseline till the end of the primary window (=duration of LISA administration + 15 minutes after removal of the thin catheter). Mean values of crSO2 during the 5min before intervention started is defined as the baseline. crSO2 parameters with beginning five minute before surfactant administration till 15 minutes after extubating will be assessed every minute.

SECONDARY OUTCOMES:
Change in arterial oxygen saturation (SpO₂) during and after LISA | From baseline (= 5min before insertion of the LISA catheter) till 15 minutes after removal of the thin catheter
  The secondary outcome measure will be the maximum change of SpO2 from baseline till the end of the primary window (=duration of LISA administration + 15 minutes after removal of the thin catheter). Mean values of SpO2 during the 5min before intervention started is defined as the baseline. SpO2 parameters with beginning five minute before surfactant administration till 15 minutes after extubating will be assessed every minute.
Change in heart rate (HR) during and after LISA | From baseline (= 5min before insertion of the LISA catheter) till 15 minutes after removal of the thin catheter
  The secondary outcome measure will be the maximum change of HR from baseline till the end of the primary window (=duration of LISA administration + 15 minutes after removal of the thin catheter). Mean values of HR during the 5min before intervention started is defined as the baseline. HR parameters with beginning five minute before surfactant administration till 15 minutes after extubating will be assessed every minute.
Change in crSO2 up to three hours after LISA | Beginning of the surfactant administration (insertion of the thin catheter) till three hours after LISA procedure
  The secondary outcome measures will be crSO2 up to three hours after surfactant administration defined as maximum changes/drop from starting with the beginning of the surfactant administration after insertion of the thin catheter till three hours after LISA procedure. Vital parameters will be assessed every five minutes till three hours after LISA procedure.
Change in SpO2 up to three hours after LISA | Beginning of the surfactant administration (insertion of the thin catheter) till three hours after LISA procedure
  The secondary outcome measures will be SpO2 up to three hours after surfactant administration defined as maximum changes/drop from starting with the beginning of the surfactant administration after insertion of the thin catheter till three hours after LISA procedure. Vital parameters will be assessed every five minutes till three hours after LISA procedure.
Change in HR up to three hours after LISA | Beginning of the surfactant administration (insertion of the thin catheter) till three hours after LISA procedure
  The secondary outcome measures will be HR up to three hours after surfactant administration defined as maximum changes/drop from starting with the beginning of the surfactant administration after insertion of the thin catheter till three hours after LISA procedure. Vital parameters will be assessed every five minutes till three hours after LISA procedure.
Change in mean arterial blood pressure (MABP) up to three hours after LISA | Beginning of the surfactant administration (insertion of the thin catheter) till three hours after LISA procedure
  The secondary outcome measures will be MABP up to three hours after surfactant administration defined as maximum changes/drop from starting with the beginning of the surfactant administration after insertion of the thin catheter till three hours after LISA procedure. Vital parameters will be assessed every five minutes till three hours after LISA procedure.
Amount of bradycardia | Beginning of the surfactant administration (insertion of the thin catheter) till three hours after LISA procedure
  The secondary outcome measure will be the amount of bradycardia (in minutes) up to three hours after surfactant administration
Amount of cerebral hypoxia | Beginning of the surfactant administration (insertion of the thin catheter) till three hours after LISA procedure
  The secondary outcome measure will be the amount of cerebral hypoxia (in minutes) up to three hours after surfactant administration
Amount of systemic hypoxia | Beginning of the surfactant administration (insertion of the thin catheter) till three hours after LISA procedure
  The secondary outcome measure will be the amount of systemic hypoxia (in minutes) up to three hours after surfactant administration
Amount of supplemental oxygen | Beginning of the surfactant administration (insertion of the thin catheter) till three hours after LISA procedure
  The secondary outcome measure will be the amount of supplemental oxygen up to three hours after surfactant administration
Need for repeat surfactant administraiton | Within 48 hours after first LISA procedure
  Proportion of infants requiring a second surfactant dose as per clinical indication.
Need for invasive ventilation | Within 48 hours after first LISA procedure
  Proportion of infants requiring intubation and mechanical ventilation due to respiratory failure.
Bronchopulmonary dysplasia (BPD) | At 36 weeks corrected gestational age
  Incidence of BPD, defined as oxygen and/or respiratory support requirement at 36 weeks postmenstrual age.
Intraventricular haemorrhage (IVH) | At 40 weeks of corrected age
  Incidence of any IVH assessed by cranial ultrasound
Periventricular leukomalacia (PVL) | At 40 weeks of corrected age
  Presence of cystic PVL or increased periventricular echogenicity consistent with white matter injury.
Retinopathy of prematurity | At 40 weeks of corrected age
  Presence of ROP
Necrotizing enterocolitis (NEC) | At 40 weeks of corrected age
  Presence of NEC
Mortality | At 40 weeks of corrected age
  Occurence of mortality during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Division of Neonatology, Department of Pediatrics and Adolescent Medicine, Graz, Austria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study population consists of extremely preterm neonates, and complete anonymisation cannot be guaranteed due to the small sample size and highly specific physiological datasets (continuous cerebral and systemic oxygenation monitoring).
  Sharing such detailed physiological and clinical data could potentially allow re-identification of individual participants, even after de-identification.
  In addition, the national ethics approval and parental consent cover data use exclusively for the present research project and associated publications, not for open data sharing.
  Aggregated and summarised results will, however, be made publicly available through peer-reviewed publications and trial registries upon study completion.